CLINICAL TRIAL: NCT06091150
Title: Endovascular Management of Direct Carotid-cavernous Fistula
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Tharwat, Resident physician, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-9-10MS
Record Dates: First submitted 2023-09-30; First posted 2023-10-19 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Carotid-Cavernous Sinus Fistula
MeSH Terms: conditions — Carotid-Cavernous Sinus Fistula

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with direct carotid cavernous fistula (Experimental): Endovascular management using coils , detachable balloons or embolizing agents
  Interventions: Procedure: Endovascular management of direct carotid-cavernous fistula

INTERVENTIONS:
Procedure: Endovascular management of direct carotid-cavernous fistula — Coiling and embolization of direct carotid-cavernous fistula

SUMMARY:
Carotid-cavernous fistula (CCF) refers to an aberrant arteriovenous communication between the carotid arterial system and the venous compartments of the cavernous sinus (CS) Direct CCFs are when there is a direct fistulous connection between the cavernous sinus and cavernous segment of the internal carotid artery (ICA), it is called direct or type-A CCF and occur secondary to a traumatic tear in the artery from a skull base fracture, from the acceleration-deceleration force of a traumatic injury, or from an iatrogenic injury following an endovascular intervention or a trans-sphenoidal procedure. They can also occur spontaneously following an ICA aneurysm rupture or weakening of the arteries from a genetic condition with subsequent development of chemosis, proptosis, bruit, headache, and/or gradual decrease in vision either unilaterally or bilaterally. High incidence of motor car accidents in Egypt carries a relative high incidence of carotid cavernous fistula. Since direct (type A) CCFs are high flow fistulas with acute/ subacute presentation and may cause serious complications, such as permanent vision loss or intracranial hemorrhage, they have to be treated early. CT orbit and MRI often help to confirm the initial diagnosis of CCF demonstrating extraoccularmuscleenlargement,dilatationofoneorbothsuperiorophthalmic veins and enlargement of the affected cavernous sinus.Because of its high spatial and temporal resolution ; the gold standard for evaluation of CCF is digital subtraction angiography; but currently CT angiography is the non invasive modality of choice for its evaluation .Previously surgical intervention included suturing or clipping the fistula, packing the cavernous sinus or ligating the internal carotid artery procedures .Currently endovascular management is the main stay of treatment for patients that fail or not suitable for conservative management and compression therapy. Significant advances in stent and catheter design now make it possible in many instances to deploy covered stents , detachable balloons, detachable coils, both detachable balloons and coils , both detachable and push coils , parent arterial occlusion and using of embolizing materials depending on availability, patient's affordability, type of fistula, and ease of use.Trans femoral catheterization is the main approach. However, trans-radial approach will be considered in patients with advanced iliofemoral diseases

ELIGIBILITY:
Inclusion Criteria:

* Patients with direct type of carotid cavernous fistula

Exclusion Criteria:

* End stage renal disease
* haemodynamically unstable patients.
* Patients with impaired coagulation profile.

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Change in patient proptosis as measured by millimeters after endovascular interventional procedures | 6 months
  Change in patient proptosis measured in millimeters by ruler's test and by plain CT orbit after endovascular management and comparison with the degree of pre-procedural patient proptosis measured in millimeters .
Change in patient visual acuity as assessed by Snellen chart | 6 months
  Change in patient visual acuity assessed by Snellen chart and its comparison with patient pre-procedural vison acuity assessed by Snellen chart.

SECONDARY OUTCOMES:
Assessment of post-procedural change in superior ophthalmic vein caliber measured in millimeters | 6 months
  Change in the caliber of superior ophthalmic vein in millimeters and comparison with the contralateral symptom free side and its comparison with pre-procedural superior ophthalmic vein congestion measured in millimeters .

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmad Tharwat, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All study and its results will be allowed in my institute website